CLINICAL TRIAL: NCT01277575
Title: Multicenter Study of Non-invasive Repetitive Paraorbital Alternating Current Stimulation of the Brain: Therapy for Aphasy
Brief Title: Non-invasive Repetitive Paraorbital Alternating Current Stimulation Therapy for Aphasia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: recruitment efforts did not result in a sufficient number of patients
Sponsor: University of Magdeburg (Other)
Collaborators: EBS Technologies GmbH (Industry)
Responsible Party: Dr. Ephrat Lahmer-Naim, Clinical Trials Manager, EBS Technologies GmbH
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EBS-PP-2010-08-25-001
Record Dates: First submitted 2011-01-14; First posted 2011-01-17 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2011-01

CONDITIONS: Aphasia
Keywords: stroke; aphasia; language
MeSH Terms: conditions — Aphasia; Stroke; Language

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Verum stimulation (Experimental): repetitive transorbital alternating current stimulation (rtACS)
  Interventions: Device: rtACS stimulation (Verum condition)
- Placebo stimulation (Sham Comparator): Sham stimulation (placebo condition) no intervention
  Interventions: Device: placebo condition

INTERVENTIONS:
Device: rtACS stimulation (Verum condition) — Repetitive, transorbital alternating current stimulation (rtACS) is applied with multi-channel device generating weak current pulses in predetermined firing bursts of 2 to 9 pulses. The amplitude of each current pulse is below 1000 microA. Current intensity is individually adjusted according to how well patients perceived phosphenes, i.e. any sensation of flickering light in response to the rtACS stimulation
  Arms: Verum stimulation
Device: placebo condition — A clicking sound is presented and the same electrode montage set-up is used during rtASC- and Placebo-stimulation, except that placebo patients received no current (stimulator turned off).
  Arms: Placebo stimulation

SUMMARY:
The investigators assess if repetitive, transcranial alternating current stimulation (rtACS) can improve the speaking quality of the aphasic patient as well as other communication skills as naming, repeating and understanding spoken words, reading and writing. Further, it will be assessed if memory and attentiveness deficiencies after 10 days of therapy with brain stimulation are stabilized and remain stable after a training-free period of 60 days.

ELIGIBILITY:
Inclusion Criteria:

* stroke
* lesion age at least 6 months
* aphasia with at least moderate severity according to Aachener Aphasia Test (AAT)
* age between 40 and 75
* German-speaking (at a native speaking level)

Exclusion Criteria:

* cognitive or speech-language therapy during the 2-weeks stimulation course
* intensive language training when exceeding 1 hour, 2 times a week during the 2-weeks stimulation course and the follow-up period (60 days after stimulation was completed)
* additional neurological diseases, e.g. surgical brain tumor removal, untreated tumor disease, acute traumatic brain injury, and/or craniotomy
* (severe) dysarthria
* untreated hypertension exceeding 160/100 mmHg (patients with treated hypertension and blood pressure below 160/100 mmHg can be included)
* increased risk of vascular thrombosis
* epilepsy, photo sensitivity, acute focal findings (patients without focal findings or epileptiform discharges can be included when they had only a single seizure more than 10 years ago)
* dementias and neurodegenerative diseases
* significant psychiatric disturbances, e.g. schizophrenia
* major attention and/or memory deficits
* major hearing loss
* patients with uncorrected visual deficits
* severe global aphasia
* modality-specific disorders (pure speech apraxia, pure alexia, pure agraphia)
* electric or electronic implants (e.g. heart pacemakers)
* metal artefacts located at the head
* medication with impact on the central nervous system (e.g. antidepressant or sedative drugs)
* participation in another trial
* pregnant or breastfeeding women

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
improvement of speaking | between baseline and 60 days after stimulation
  assessed by the following tests:
  * Expressive speaking: ANELT (Amsterdam Nijmegen Everyday Language Test), Aachener Aphasie Test
  * receptive speaking: ANELT (Amsterdam Nijmegen Everyday Language Test), Aachener Aphasie Test

SECONDARY OUTCOMES:
successful stabilization of language | 60 days after stimulation
speaking functions 1 - communicative skills | baseline to 60 days after stimulation
  * reading and writing: Aachener Aphasy Test
  * attentiveness: TAP test battery
  * working Memory: Wechsler Memory scale-Revised (WMS-R)
  * emitional state: Vision Analogous Mood Scale (VAMS)
speaking functions 2 - spontaneous speech faculty | baseline to 60 days after stimulation
  * reading and writing: Aachener Aphasy Test
  * attentiveness: TAP test battery
  * working Memory: Wechsler Memory scale-Revised (WMS-R)
  * emitional state: Vision Analogous Mood Scale (VAMS)
speaking functions 3 - naming | baseline to 60 days after stimulation
  * reading and writing: Aachener Aphasy Test
  * attentiveness: TAP test battery
  * working Memory: Wechsler Memory scale-Revised (WMS-R)
  * emitional state: Vision Analogous Mood Scale (VAMS)
speaking functions 4 - repeating | baseline to 60 days after stimulation
  * reading and writing: Aachener Aphasy Test
  * attentiveness: TAP test battery
  * working Memory: Wechsler Memory scale-Revised (WMS-R)
  * emitional state: Vision Analogous Mood Scale (VAMS)
speaking functions 5 - understanding | baseline to 60 days after stimulation
  * reading and writing: Aachener Aphasy Test
  * attentiveness: TAP test battery
  * working Memory: Wechsler Memory scale-Revised (WMS-R)
  * emitional state: Vision Analogous Mood Scale (VAMS)

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard A Sabel, Prof. Dr., Principal Investigator — University of Magdeburg
Locations (3):
- Germany (3):
  - Neurologische Klinik, Medizinische Fakultät der RWTH Aachen, Pauwelsstr. 30, Aachen
  - Neurologische Klinik, Brandenburg Klinik Bernau, Brandenburgallee 1, Bernau Waldsiedlung
  - Institut für Medizinische Psychologie, Leipziger Str. 44, Magdeburg